CLINICAL TRIAL: NCT06754046
Title: BELIEVE Trial: Bulking vErsus sLing for Treating Stress Urinary IncontinEnce at the Time of Vaginal prolapsE Repair
Brief Title: BELIEVE Trial: Bulking vErsus sLing for Treating Stress Urinary IncontinEnce at the Time of Vaginal prolapsE Repair (BELIEVE)
Acronym: BELIEVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Kaiser Permanente (Other); Duke University (Other); Patient-Centered Outcomes Research Institute (Other); University of California, San Diego (Other); University of California, Irvine (Other); MetroHealth Medical Center (Other); Ohio State University (Other); Northwestern University (Other); University of New Mexico (Other); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, David Sheyn, Associate professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20241497
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Stress Urinary Incontinence; Vaginal Prolapse
Keywords: midurethral sling; bulkamide; polyacrylamide hydrogel; urethral bulking; retropubic sling
MeSH Terms: conditions — Urinary Incontinence, Stress; Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Retropubic Midurethral Sling (RP-MUS) (Active Comparator): A minimally invasive surgical procedure that treats stress urinary incontinence (SUI) in women by placing a small strip of tape passed through the retropubic space, with entry and exit points in the lower abdomen or groin.
  Interventions: Device: RP-MUS
- Urethral Bulking with polyacrylamide hydrogel (PAHG) (Active Comparator): PAHG will be performed using the standard 2 mL dose injection order and number will be at the discretion of the surgeon. Patients undergoing PAHG will be given sham incisions consisting of superficial suprapubic epidermal scratches with a needle and fibrin glue at expected sling exit sites.
  Interventions: Procedure: PAHG

INTERVENTIONS:
Device: RP-MUS — a standard urethral sling placement for treatment of stress urinary incontinence
  Arms: Retropubic Midurethral Sling (RP-MUS)
Procedure: PAHG — A standard 2 mL dose injection of bulkamid (order and number will be at the discretion of the surgeon) will be given. Patients undergoing PAHG will be given sham incisions consisting of superficial suprapubic epidermal scratches with a needle and fibrin glue at expected sling exit sites.
  Arms: Urethral Bulking with polyacrylamide hydrogel (PAHG)

SUMMARY:
The goal of this clinical trial is to learn if retropubic midurethral sling (RP-MUS) or bulkamide injection (PAHG) at the time of pelvic organ prolapse repair is better from the patient's perspective. The main questions it aims to answer are:

What is the average difference in the urogenital distress inventory (UDI) long form score 24 months after surgery for each procedure? Which procedure has the fewest complications and lowest short- and long-term morbidity profile?

Participants will:

Be blinded and randomized to one of two procedures for the duration of the study, 24 months.

Complete 6 total visits for the clinical trial including validated questionnaires.

Few participants will be selected to complete a qualitative interview at 3 timepoints over 24 month duration of the study.

DETAILED DESCRIPTION:
This will be a double-blinded, non-inferiority, controlled trial utilizing a 1:1 randomization scheme to assign patients to each treatment arm (PAHG vs. RP-MUS). Patients undergoing PAHG will be given sham incisions in order to mask the type of SUI procedure they underwent. This will consist of two "earring-hole" sized superficial scratches in the epidermis and fibrin glue applied to the expected suprapubic exit sites for the RP-MUS. Sham incisions are not associated with an increased risk of infection and are considered low risk. Validated symptom questionnaires will be administered to the patient by a study investigator prior to surgery and at 1, 6, 12, and 24 months. At the final study visit, patients will be un-blinded and provided information on which SUI procedure they underwent. Unless it is necessary for subsequent care, as in the case of a procedure specific complication like a mesh erosion, patients who might require additional intervention for recurrent SUI during the study period will remain blinded to their initial treatment assignment. If patients request this information, they will be informed that they would need to exit the study, however their data would still be analyzed as part of the intention to treat protocol. Data of patients who dropout will be analyzed in the same manner. Pelvic organ prolapse procedures will be limited to native tissue repairs only and may include either or both apical and non-apical repair procedures; selection of appropriate POP repair procedure will be at the surgeon's discretion. All randomized patients will complete surveys at 12 and 24 months will assess patient recovery, satisfaction with care, and calibrating surveyed and clinically assessed outcomes to their daily life experiences. Based on prior similar studies, this number is sufficient to ensure saturation of themes83. Between 8 to 20 participants in each arm will be randomly selected from across all sites to participate in individual semi-structured telephone interviews preoperatively, at 12 months and at 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age.
* Have diagnosis of symptomatic stress urinary incontinence (SUI) as noted in their electronic health record (EHR).
* Proof of positive testing for SUI via cough stress test (CST) and/or Urodynamic (UDS) testing,
* Patients that are planning and eligible for vaginal prolapse repair and for both Retropubic Midurethral Sling (RP-MUS) and Polyacrylamide Hydrogel (PAHG)

Exclusion Criteria:

* Patients undergoing pelvic organ prolapse repair using mesh or biologic augmentation other than patient's own tissue
* Patient anticipating difficulty with completing 24-month follow-up
* Anticipation of pregnancy within subsequent 24-months or <18 months post-partum
* Hemoglobin A1c >10.0% within the past 3-months
* Current smoker > 1 pack per week
* History of neurogenic bladder
* Current use of any catheterization including but not limited to, intermittent catheterization, indwelling Foley catheter, or suprapubic catheter
* Post-void residual >150 mL felt to not be due to obstruction for prolapse
* Prior history of any anti-incontinence procedure including but not limited to any synthetic sling, fascial sling, Burch colposuspension or its variants, and urethral bulking
* Previous history of any pelvic radiation
* Patient receiving a planned concurrent procedure at the time of prolapse repair.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender assigned female at birth
Enrollment: 476 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Bothersome stress urinary incontinence symptoms as measured by urogenital distress inventory long form (UDI) | 24 months postoperatively
  a questionnaire used to assess the severity of lower urinary tract symptoms like incontinence, particularly in women, by measuring the impact of these symptoms on their quality of life. Scores range from 0 to 100, higher number indicates worse symptoms.

SECONDARY OUTCOMES:
Change in bothersome stress urinary incontinence symptoms as measured by urogenital distress inventory long form (UDI) | 1, 6 and 12 months postoperatively
  a questionnaire used to assess the severity of lower urinary tract symptoms like incontinence, particularly in women, by measuring the impact of these symptoms on their quality of life. Scores range from 0 to 100, higher number indicates worse symptoms.
Change in patient assessment of improvement as measured by the Patient Global Impression of Improvement (PGI-I) | 1 month, 6 months, 12 months and 24 months postoperatively
  Patient Global Impression of Improvement (PGI-I) score is a rating on a scale from 1 to 7 that measures a patient's perception of how their condition has changed in response to treatment
Number of retreatment for SUI as measured by medical record review/patient report | up to 24 months post operatively
Change in Lower urinary tract dysfunction research network symptom index-29 (LURN-SI-29) | preoperatively, 1, 6, 12 and 24 months postoperatively
  A patient-centric questionnaire developed to provide a comprehensive assessment of lower urinary tract symptoms including symptoms of overactive bladder and voiding dysfunction. Scoring ranges from 0 (least severe) to 100 (most severe).
Change in Female Sexual Function Inventory (FSFI) | preoperatively, 1, 6, 12 and 24 months postoperatively
  This 19 item questionnaire will assess sexual function and body image. It has a scoring range from 2 to 36 with higher scores indicating better sexual functioning.
Average of Perioperative morbidity | Up 24 months postoperatively
  Perioperative morbidity will be assessed using the Clavien-Dindo classification. The classification is a system for grading the severity of postoperative complications based on the level of intervention required to treat them. The CD classification uses five grades of severity, with Grade I being low and Grade V being death.
Pelvic organ prolapse recurrence (POP-Q) | preoperatively, 1, 6, 12 and 24 months postoperatively
  Recurrence of pelvic organ prolapse is assessed utilizing the POP-Q system classifies pelvic organ prolapse into four stages. It ranges from Stage I (most distal part of the prolapse is more than 1 cm above the hymen) to Stage IV (Complete procidentia or vault eversion)

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Cecile Ferrando, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers to ensure participant privacy is maintained and avoid any risk of invalid analyses.